CLINICAL TRIAL: NCT06117176
Title: Prospective Assessment Project of AirwaY Management-related Incidents in Adult Anaesthesia Care (PAPAYA III) - A European Multicentre Cross-sectional Observational Study
Brief Title: Prospective Assessment Project of AirwaY Management-related Incidents in Adult Anaesthesia Care PAPAYA III
Acronym: PAPAYA-III
Status: Not yet recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); University of Lausanne Hospitals (Other); Kantonsspital Aarau (Other); Charite University, Berlin, Germany (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PAPAYA III; 2023-01752 (Registry Identifier: Swissethics)
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Airway Complication of Anesthesia; Adverse Events
Keywords: Intubation, Intratracheal; Anesthesiology; Difficult Airway; Critical events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall objective of the study is to evaluate and analyze major and minor incidents during airway management in adults under anaesthesia care at all study sites. The patient characteristics, type of airway management is recorded and if airway management-related incidents occur, they are analyzed in more detail to improve patient safety in the future.

DETAILED DESCRIPTION:
It is a prospective observational cross-sectional European multi-centre study collecting health-related patient data on anaesthetic airway management over three months. This detects the incidence and nature of local airway management problems and assesses how they are solved. This will enable the investigators to identify generalisable interventions and recommendations to further improve patients' airway management to improve patient safety. During the observational period, the anaesthesia staff in charge will fill out a screening questionnaire for airway management for every patient undergoing anaesthesia care with airway management. The investigators will extract the characteristics from the local anaesthesia record system for all patients. If no event arises, there are no further requirements. If an event occurs, the anaesthesia provider will fill out an additional form asking for more details on what happened.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients requiring airway management under anaesthesia care for elective, semi-elective, urgent or emergency diagnostic procedures or interventions. Airway management includes awake and asleep tracheal intubation, insertion of supraglottic airway devices, and face mask ventilation.
* Patients older than 18 years of age
* Informed consent given or general consent in place, according to local ethics committee requirements.

Exclusion Criteria:

* Refusal to give consent or withdrawal of consent.
* Patients <18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (<18 years of age) that undergo in-hospital airway management under anaesthesia care who do not object to the use of their data collected for the purpose of this study.
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Number of airway management related incidents | 30 days
  Primary study outcome is the number of anaesthesia cases with at least one airway management related incidents in adult patients under anaesthesia care.

SECONDARY OUTCOMES:
The Incidences of the individual major incidents | 30 days
  Secondary study outcome parameters are the incidences of the major critical events and the number of incidents per case incidents.
The Incidences of the individual minor incidents | 30 days
  Secondary study outcome parameters are the incidences of the minor critical events and the number of incidents per case incidents.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Greif, MD, Prof, Study Chair — Department of Anaesthesiology and Pain Medicine, Inselspital, Bern University
Locations (4):
- Germany (2):
  - Deutsches Herzzentrum der Charité and Charité, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - CHUV Centre Hospitalier Universitaire Vaudois, Lausanne

IPD SHARING:
Plan to Share IPD: No